CLINICAL TRIAL: NCT03082313
Title: Movement-based Intervention to Promote Positive Neurodevelopmental Outcomes in Infants at Risk for Developmental Delay
Brief Title: Movement-based Infant Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Beth A. Smith, Assistant Professor of Research, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-16-00959
Record Dates: First submitted 2017-03-03; First posted 2017-03-17 (Actual); Results first posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-02

CONDITIONS: Infant Development; Infant,Premature; Infant, Very Low Birth Weight; Infant, Small for Gestational Age; Infant Conditions
Keywords: infant; leg movement; wearable sensors; early intervention
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Movement intervention (Experimental): The intervention promotes movement experience from 3 months to sitting onset in infants at risk for developmental delay (AR). The goal of the intervention is to increase amount and type of infant leg movement experience above 1200 movements per hour of awake time.
  Interventions: Behavioral: Movement Intervention

INTERVENTIONS:
Behavioral: Movement Intervention — At each visit, the caregiver will be reminded of the infant's movement rate from the last visit. The research team will help the caregiver to determine possible ways to achieve the goal of 1200 movements per hour of awake time. Strategies to increase leg movements will be encouraged based on the infant's developmental level and what they demonstrate a response to, including: shake a toy when infant moves legs, sing a line of a song when infant moves legs, change the position of the infant to encourage more leg movement, or lightly tickle the legs and feet of the infant. The intervention will be based upon the GAME (Goals - Activity - Motor Enrichment) protocol, a motor learning, environmental enrichment intervention that has recently been shown to be effective for improving motor skills in infants at high risk of cerebral palsy compared to standard care.

SUMMARY:
The objective is to pilot test the effectiveness of an evidence-based intervention to promote positive neurodevelopmental outcomes in infants at risk for developmental delay. The intervention promotes movement experience from 3 months to sitting onset.

DETAILED DESCRIPTION:
Aim: Our purpose was to assess daily leg movement rate before and after a caregiver-provided in-home intervention for infants at risk for developmental disability. We also assessed adherence and quality of caregiver-child interaction.

Methods: Twelve infants, at risk for developmental disabilities, and their caregivers participated in an intervention focused on increasing leg movements. Intervention started between 3- and 6-months cor- rected age and ended once the infant was able to sit independently or at 9 months corrected age, whichever occurred first. Infants were assessed monthly.

ELIGIBILITY:
Inclusion Criteria:

* Infants will be 3 months of adjusted age at the first visit, +/- 10 days. Infants will be defined as at risk if they qualify for high risk infant follow up care as defined by California Children's Services.

Exclusion Criteria:

* Infants with congenital malformations of the legs will be excluded.

Ages: 3 Months to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth A Smith, PT, PhD, Principal Investigator — University of Southern California
Locations (1):
- Infant Neuromotor Control Laboratory, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Movement Intervention
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Movement Intervention
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 12
leg movement rate [Median (Full Range); unit: average leg movements per hour awake] | 1294 [506 to 2105]

OUTCOME MEASURES:

1. Primary Outcome: Movement Rate
Description: leg movements produced per hour of awake time, assessed using wearable sensors
Time Frame: post intervention (intervention duration ranged from 2-6 months)
Population: all infants enrolled in the study
Measure: Median (Full Range); unit: average leg movements per hour awake
Arm/Group | Movement Intervention
Number analyzed (Participants) | 12
average leg movements per hour awake | 1278 [655 to 2078]

ADVERSE EVENTS:
Time Frame: across the duration of each infants' participation (range 2-6 months)
Arm/Group | Movement Intervention
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT03082313/Prot_SAP_000.pdf